CLINICAL TRIAL: NCT01017172
Title: Safety and Immune Response to Adjuvanted A(H1N1)v Influenza Vaccine in HIV-1 Infected and Immunosuppressed Adults
Brief Title: Safety and Immune Response to Adjuvanted A(H1N1)v Influenza Vaccine in HIV-1 Infected and Immunosuppressed Adult Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Collaborators: HIVCENTER (Unknown)
Responsible Party: Markus Bickel / MD, HIVCENTER, JW Goethe University Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JWG11.2009
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: HIV-1 Infection; Cancer; Immunosuppression
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: serologic testing — Serologic testing will be performed baseline, day 21 and day 42

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of an adjuvanted A(H1N1)v influenza vaccine in HIV-infected and immunosuppressed patients after one and two injections.

DETAILED DESCRIPTION:
The efficacy of an adjuvanted A(H1N1)v influenza vaccine in HIV-infected and immunosuppressed patients is unknown. Therefore we aim to investigate the immunoresponse as assessed by a anti-hemagglutinin assay before, 21 days after the first and 21 days after the second vaccination. The safety of the vaccination will be recorded by a standardized questionaire.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age >18
* HIV-1 infection
* cancer
* immunosuppressive treatment

Exclusion Criteria:

* not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To investigate the immunogenicity via anti-hemagglutinin responses following an adjuvanted H1N1 vaccination in HIV-positive and immunosuppressed adult patients | baseline, day 21, day 42

SECONDARY OUTCOMES:
To evaluate the effect of pre-existing anti-influenza immunity and recent history of seasonal influenza and H5N1 vaccination on seroresponses to the H1N1 influenza vaccine | baseline
To evaluate potential adverse reactions of the H1N1 vaccine | baseline, day 21, day 42

CONTACTS AND LOCATIONS:
Overall Officials: Markus Bickel, MD, Study Director — JW Goethe University Clinic; Christoph Stephan, MD, Study Chair — JW Goethe University Clinic; Hans R Brodt, MD, Principal Investigator — JW Goethe University Clinic
Locations (1):
- Hivcenter, Frankfurt, Germany

REFERENCES:
- [Derived] Bickel M, Lassmann C, Wieters I, Doerr HW, Herrmann E, Wicker S, Brodt HR, Stephan C, Allwinn R, Jung O. Immune response after a single dose of the 2010/11 trivalent, seasonal influenza vaccine in HIV-1-infected patients and healthy controls. HIV Clin Trials. 2013 Jul-Aug;14(4):175-81. doi: 10.1310/hct1404-175. PMID 23924590
- [Derived] Gueller S, Allwinn R, Mousset S, Martin H, Wieters I, Herrmann E, Serve H, Bickel M, Bug G. Enhanced immune response after a second dose of an AS03-adjuvanted H1N1 influenza A vaccine in patients after hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2011 Oct;17(10):1546-50. doi: 10.1016/j.bbmt.2011.02.004. Epub 2011 Feb 13. PMID 21324375
- [Derived] Bickel M, von Hentig N, Wieters I, Khaykin P, Nisius G, Haberl A, Stephan C, Herrmann E, Doerr HW, Brodt HR, Allwinn R. Immune response after two doses of the novel split virion, adjuvanted pandemic H1N1 influenza A vaccine in HIV-1-infected patients. Clin Infect Dis. 2011 Jan 1;52(1):122-7. doi: 10.1093/cid/ciq003. PMID 21148530
- [Derived] Bickel M, Wieters I, Khaykin P, Nisius G, Haberl A, Stephan C, Von Hentig N, Herrmann E, Doerr HW, Brodt HR, Allwinn R. Low rate of seroconversion after vaccination with a split virion, adjuvanted pandemic H1N1 influenza vaccine in HIV-1-infected patients. AIDS. 2010 Jun 1;24(9):F31-5. doi: 10.1097/QAD.0b013e3283398da1. PMID 20559034